CLINICAL TRIAL: NCT02037178
Title: Screening for Arteriopathy in General Medicine: a Preliminary Feasibility Study
Acronym: DAG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/JLLD-01; 2013-A01583-42 (Other: RCB number)
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Obliterative Arteriopathy
Keywords: Peripheral Obliterative Arteriopathy of the legs; Screening by generalists; Ultrasound
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: See inclusion/exclusion criteria.
  Intervention: First ultrasound reading
  Intervention: Second ultrasound interpretation
  Interventions: Other: First ultrasound reading; Other: Second ultrasound interpretation

INTERVENTIONS:
Other: First ultrasound reading — First ultrasound reading of the sub-renal abdominal aorta by a general practitioner.
Other: Second ultrasound interpretation — The untrasound images recorded by general practitioners will be interpreted a second time by an expert in vascular medecine, and evaluated for their image quality.

SUMMARY:
The main objective of this study is to evaluate the inter-observer concordance when measuring the maximum value of the external antero-posterior diameter of the sub-renal aorta (both cross-sectional and longitudinal ultrasound views are measured). The first measure is made by a general practitioner in private practice; second reading are made by an expert in vascular medicine.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To assess the prevalence of Abdominal Aortic Aneurysm (AAA) detected by ultrasound measurement of the anterior and posterior longitudinal outer diameter of the sub-renal abdominal aorta in a high cardiovascular risk population consulting with general practitioners (defined according to recommendations stated by the French Society of Vascular Medicine).

B. To assess the prevalence of Peripheral Obliterative Arteriopathy of the Legs (POAL) by measuring the Systolic Pressure Index (SPI) at the toe (ratio of arterial pressure in upper limbs versus lower limbs). Measures are made by a general practitioner in the same population.

C. To assess the quality and interpretability of ultrasound recordings and ultrasound acquistion failure rate. These second measures are made by an expert in vascular medecine. This evaluation with use a 3-level scale:

1. appropriate image was not obtained or not recognized expert - uninterpretable
2. poor image quality - interpretable
3. image of good or very good quality - interpretable

D. To calculate the impact of risk cofactors such as hypertension , smoking, age and family history among patients diagnosed with AAA.

E. Evaluation of general practitioner training from a qualitative and quantitative point of view after 4 h of training organized by Dr. Bobbià .

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient falls into one of the following 4 groups as defined by the French Society of Vascular Medecin (2006):
* (1) Men and women 60-75 years of age who are active smokers or ex-smokers
* (2) Men over 75 years of age
* (3) Women over 75 years of age who smoke and who have known hypertension
* (4) Men and women over 50 years of age with a family history of aneurysm of the abdominal aorta

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject has an allergy to the gel used for ultrasound examination.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations consists of men and women consulting with general practitioners and who are at high risk for cardio vascular disease a defined by the French Society of Vascular Medecin.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Largest external antero-posterior diameter of the sub-renal abdominal aorta (mm) | Baseline (day 0)
  Measures made using both cross-sectional and longitudinal ultrasounds.

SECONDARY OUTCOMES:
SPI at the toe (mmHg) | baseline (Day 0)
Largest external antero-posterior diameter of the sub-renal abdominal aorta (mm) : second interpretation of echographic material by a second expert | maximum of three months
  Measures made using both cross-sectional and longitudinal ultrasounds.
Ultrasound quality as assessed by the second expert | maximum of three months
  This evaluation with use a 3-level scale:
  1. appropriate image was not obtained or not recognized expert - uninterpretable
  2. poor image quality - interpretable
  3. image of good or very good quality - interpretable

OTHER OUTCOMES:
Age | baseline (day 0)
Smoker? yes/no | baseline (day 0)
Hypertension? yes/no | baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: David Costa, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Centre Médico Sportif, Nîmes